CLINICAL TRIAL: NCT06695416
Title: Community-based Partnership's Efficacy in Decreasing Injury Rates At Night in Dallas, TX
Status: Recruiting | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 003.TRA.2023.D
Record Dates: First submitted 2023-07-06; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-07

CONDITIONS: Blood Alcohol Concentration; Drunk Driving
MeSH Terms: conditions — Driving Under the Influence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
According to the Centers for Disease Control and Prevention (CDC), "88,000 people die every year due to alcohol-related issues including homicide, sexual assault, intimate partner violence, and suicide". In the city of Dallas, violent crimes have decreased by roughly 4% in 2022 compared to 2021. Dallas Police Department (DPD) implemented changes in May 2021 to combat violent crimes.

DETAILED DESCRIPTION:
To address these issues, 24Hour Dallas, a community-based non-profit organization, has utilized public health approaches at the business and city level. Their overarching goals are to reduce drunk driving, violence against women, human trafficking, and general violence or injuries related to alcohol use, all within the nighttime hours of 6pm and 6am through the application of their Good Neighbor initiative and Copper Star certification for businesses. Both the Good Neighbor initiative and the Copper Star certification follow a model from Safe Night LLC, an organization that was built on the premise of The Arlington Restaurant Initiative in Arlington, Virginia.

ELIGIBILITY:
Inclusion Criteria:

* • Chief complaint or diagnosis associated with a trauma mechanism of injury: assault (i.e., gunshot wounds, knife wounds, general assault, or sexual assault), MVC, motorcycle/all-terrain vehicle collision (MCC), or auto-ped/bicycle collision

  * Injury occurred between 6pm-6am
  * Injury occurred in City of Dallas, TX

Exclusion Criteria:

* • Injuries from mechanism other than assault, MVC, MCC, or auto-ped/bicycle

  * Assault occurs outside of 6pm-6am window
  * Assault occurred outside of Dallas city limits

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chief complaint or diagnosis associated with a trauma mechanism of injury: assault (i.e., gunshot wounds, knife wounds, general assault, or sexual assault), MVC, motorcycle/all-terrain vehicle collision (MCC), or auto-ped/bicycle collision
  * Injury occurred between 6pm-6am
  * Injury occurred in City of Dallas, TX
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-04-28 (Actual); Primary Completion 2025-04-28 (Estimated); Study Completion 2025-04-28 (Estimated)

PRIMARY OUTCOMES:
Number of ED visits with implementation of 24HourDallas Copper Star Certification | 12 hours
  Number of ED visits that are associated with a mechanism of injury of assault or MVC with either a positive BAC level or a positive Audit C screen between 6pm and 6am before and after implementation of 24HourDallas Copper Star Certification in Dallas.
Number of Sexual Assault with implementation of Copper Star Certification in Dallas | 12 hours
  Number of Sexual Assault Nurse Examiner (SANE) examinations done between 6pm and 6am before and after implementation of Copper Star Certification in Dallas.
Number of ED Visits caused by Assault Injuries | 12 hours
  Number of ED Visits by females with a chief complaint of diagnosis associated with a mechanism of injury related to assault
Number of human trafficking cases with implementation of Copper Star Certification in Dallas | 12 hours
  Number of human trafficking cases between 6pm and 6am before and after implementation of Copper Star Certification in Dallas.

SECONDARY OUTCOMES:
Location of assaults | 12 hours
  Locations of assaults between 6pm-6am
  * Mechanism of injury of assaults between 6pm-6am
  * Injury rates between 6pm-6am
  * Mortality rates between 6pm-6am

CONTACTS AND LOCATIONS:
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States